CLINICAL TRIAL: NCT04598308
Title: EUROpean Coronary microCirculatory Resistance and Absolute Flow Trial: An European Registry
Brief Title: EUROpean Coronary microCirculatory Resistance and Absolute Flow Trial
Acronym: EURO-ccraft
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Onze Lieve Vrouwziekenhuis Aalst (Other)
Responsible Party: Principal Investigator, Danielle Keulards, Principal investigator, Catharina Ziekenhuis Eindhoven
Other Study IDs: NL74650.100.20
Record Dates: First submitted 2020-10-09; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Microvascular Angina; Microvascular Coronary Artery Disease; Coronary Vasospasm; Microvascular Resistance
Keywords: coronary microvascular disease; ANOCA; epicardial spasm
MeSH Terms: conditions — Microvascular Angina; Coronary Vasospasm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing invasive assessment of the microcirculation: All patients are eligible for participation in this registry if they are undergoing coronary angiography with or without coronary intervention for any reason and if an indication for the foreseen intracoronary physiologic measurements is present according to the discretion of the investigating operator. There are no specific exclusion criteria other than contraindications for physiologic measurements in general.
  Interventions: Diagnostic Test: absolute flow and resistance measurements

INTERVENTIONS:
Diagnostic Test: absolute flow and resistance measurements — This registry only collects all measurement data from normal/routine physiologic assessment in the cathlab. These measurements are performed on a daily basis
  Short description of the procedure Coronary angiography, PCI (if indicated), and physiologic measurements are performed completely according to normal routine. Physiologic measurements may include FFR, NHPR, IMR, CFR, absolute flow (Q) and microcirculatory resistance (Rmicro or MRR) measurement.
  Intention to measure Q and Rmicro are mandatory to be included in this registry.
  Use of drugs either during or after the procedure should also exactly identical to normal routine.

SUMMARY:
Rationale: coronary microvascular disease is a relatively 'new' entity within the field of cardiology. The investigators are able to investigate the microcirculation by measurements performed in the catheterization laboratory. But even though measurements are performed on a daily basis, a lot of questions regarding microvascular disease remain. The rationale of this registry is to get an overview of patients and measurement values in daily routine practice.

Objective and main endpoint: No previous registries have been set-up where coronary blood flow and resistance was systematically stored. Therefore the analyses will be mainly descriptive. The objective is to acquire a better insight in the indications and use of this technique in everyday practice , its consequences for clinical decision making, and to enable interventionalists to exchange mutual knowledge about this specific methodology and about the coronary microcirculation in general.

Study design: prospective registry

Study population: All patients who underwent coronary angiography with or without coronary intervention for any reason and if an indication for the foreseen intracoronary physiologic measurements is present according to the discretion of the operator.

Intervention (if applicable): none, only usage of measurement data. The only 'intervention' for all patients is a questionnaire.

DETAILED DESCRIPTION:
This registry only collects all measurement data from normal/routine physiologic assessment in the cathlab. These measurements are performed on a daily basis. The following paragraph will explain these routine measurements briefly.

Short description of the procedure Coronary angiography, PCI (if indicated), and physiologic measurements are performed completely according to normal routine. Physiologic measurements may include FFR, NHPR, IMR, CFR, absolute flow (Q) and microcirculatory resistance (Rmicro or MRR) measurement.

Intention to measure Q and Rmicro are mandatory to be included in this registry.

If there is failure to measure Q and/or Rmicro , it should be carefully noted including the reason for failure.

Coronary physiologic measurements may be performed either prior or after PCI, if applicable. If they are performed before PCI, it is recommended (according to Good Clinical Practice) but not absolutely mandatory to repeat these measurements also after PCI.

As said, the invasive procedure itself, including all measurements, should be performed completely according to clinical routine. Use of drugs either during or after the procedure should also exactly identical to normal routine.

ELIGIBILITY:
Inclusion criteria:

* All patients are eligible for participation in this registry if they are undergoing coronary angiography with or without coronary intervention for any reason and if an indication for the foreseen intracoronary physiologic measurements is present according to the discretion of the investigating operator.
* >18 and <90 years of age
* able to give informed consent

Exclusion criteria:

- There are no specific exclusion criteria other than contraindications for physiologic measurements in general.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: see above
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
clinical treatment assessment | 1 year
  change in clinical decision making after invasive assessment of the microcirculation

SECONDARY OUTCOMES:
IMR and resistance measurement | 2 years
  comparison between IMR and microvascular R measurements in WU

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided